CLINICAL TRIAL: NCT00209313
Title: A Randomized, Double-blind, Placebo-controlled Crossover Trial of Acyclovir for Suppression of HSV and HIV Shedding in HIV-1, HSV-2 Coinfected Persons in Cameroon
Brief Title: Usage of Acyclovir for Suppression of HIV-1 and HSV-2 Coinfected Persons in Cameroon
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Institute for the Development of Africa (Unknown)
Responsible Party: Anna Wald, MD, MPH, Fred Hutchinson Cancer Research Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: IR File 5687; AI 30731 (Project 1)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-12-16 (Estimated); Status verified 2011-12

CONDITIONS: HIV-1 and HSV-2 Coinfection; HIV Infections
Keywords: HIV-1; HSV-2; Coinfection; Africa; Cameroon
MeSH Terms: conditions — HIV Infections; Coinfection | interventions — Acyclovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Acyclovir 800 mg twice daily for 8 weeks, two week washout, 8 weeks placebo
  Interventions: Drug: Acyclovir
- 2 (Other): 8 weeks placebo, 2 week washout, 8 weeks 800 mg acyclovir twice daily
  Interventions: Drug: Acyclovir

INTERVENTIONS:
Drug: Acyclovir — Acyclovir 800 mg twice daily or placebo

SUMMARY:
The study proposed that both clinical and subclinical HSV reactivation is associated with increased HIV shedding from mucosal surfaces, which may increase the infectiousness of HIV-1/HSV-2 coinfected persons. To test this hypothesis, we will control HSV reactivation with acyclovir, a safe medication that is proven to reduce HSV shedding, and measure HIV levels in blood, genital, and pharyngeal secretions. The study hypothesizes that acyclovir will reduce HIV shedding from mucosal surfaces of HIV-1/HSV-2 coinfected individuals.

DETAILED DESCRIPTION:
The main objective is to assess the reduction in genital HIV-1 shedding associated with daily acyclovir for suppression of HSV-2 reactivation.

All patients will be treated with the usual antibiotic treatment for any sexually transmitted infections that are diagnosed during the study. In addition, half will receive acyclovir for 8 weeks , whilst the other half will receive a placebo for 8 weeks. The study medication will reverse in the second 8 weeks of the study. The patients will attend the clinic 3 times per week during the first and the last 8 weeks of the study and once every week during the washout period in the middle of the study - for a total of 18 weeks per participant. At each visit genital and oral samples will be collected. A blood sample will also be collected. For women participants, pregnancy test will be performed. The clinic will provide both pre- and post-HIV test counseling.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and above
* Documented HIV-seropositive
* HSV-2 seropositive as determined by Focus EIA
* Not intending to move out of the area for the duration of study participation
* Willing and able to:

  1. provide independent written informed consent
  2. undergo clinical evaluations
  3. take study drug as directed
  4. adhere to follow-up schedule
* Bacterial STDs (symptomatic STD syndromes or laboratory-confirmed asymptomatic gonorrhea, chlamydia, syphilis) are treated within two weeks if study enrollment and random assignment.

Exclusion Criteria:

* Women who meet any of the following criteria are not eligible for this study.

  1. Known history of adverse reaction to acyclovir
  2. Planned open label use of acyclovir, valacyclovir, or famciclovir
  3. Positive pregnancy test
  4. Active opportunistic infection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-03; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
HSV and HIV viral shedding | 18 weeks

SECONDARY OUTCOMES:
HSV suppression and HIV shedding | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Francois-Xavier Mbopi-Keou, M.Sc, PhD, Principal Investigator — Institute for the Development of Africa
Locations (1):
- Hospital Central, Yaoundé, Cameroon